CLINICAL TRIAL: NCT01859273
Title: Adherence Enhancement for Renal Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, John W. McGillicuddy, Associate Professor of Surgery, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00011702
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2016-06-10 (Estimated); Status verified 2016-06

CONDITIONS: Renal Failure; Medication Adherence; Hypertension
Keywords: renal failure; medication adherence; hypertension
MeSH Terms: conditions — Renal Insufficiency; Medication Adherence; Hypertension | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (No Intervention): Standard Care after kidney transplantation
- mHealth (Experimental): subjects provided with electronic medication tray, electronic blood pressure cuff, and a smart phone.
  Interventions: Behavioral: mHealth

INTERVENTIONS:
Behavioral: mHealth — mHealth prototype system consisting of electronic medication tray, blood pressure cuff and smart phone
  Arms: mHealth

SUMMARY:
Despite significant advances in the care of kidney transplant recipients, long term graft survival after renal transplantation remains suboptimal. Medication nonadherence and clinical inertia are key contributors to graft loss. The purpose of the proposed RCT feasibility study is to evaluate impact of a "bundled" wireless real time medication reminder system and blood pressure monitoring system in combination with a cognitive behavioral adherence skills enhancement program upon medication adherence, therapeutic drug concentration, and blood pressure, in nonadherent kidney transplant recipients with hypertension. We propose to recruit 60 kidney transplant recipients in phase 1 with 20 non-adherent continuing to phase 2 for a 5-month feasibility RCT.

ELIGIBILITY:
Inclusion Criteria:

* Persons > 21 years of age
* first time recipient of a solitary kidney transplant
* prescribed at least 3 medications for immunosuppression and hypertension
* previous history of non-adherence
* functioning kidney transplant
* ability to speak, hear and understand English
* able to use medication delivery device and self administer medications
* able to operate blood pressure monitor
* comfortable using cell phone
* no other diagnosis that might shorten lifespan
* transplant physician's assent that the patient can participate

Exclusion Criteria:

* failure to meet all inclusion criteria

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-09; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
medication adherence | 5 months
  adherence to immunosuppressive medications

SECONDARY OUTCOMES:
blood pressure | 5 months
  resting blood pressure

OTHER OUTCOMES:
acceptability | 5 months
  patients' willingness to utilize the protocol mHealth system

CONTACTS AND LOCATIONS:
Overall Officials: john w mcgillicuddy, md, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] De Geest S, Borgermans L, Gemoets H, Abraham I, Vlaminck H, Evers G, Vanrenterghem Y. Incidence, determinants, and consequences of subclinical noncompliance with immunosuppressive therapy in renal transplant recipients. Transplantation. 1995 Feb 15;59(3):340-7. PMID 7871562
- [Background] Vlaminck H, Maes B, Evers G, Verbeke G, Lerut E, Van Damme B, Vanrenterghem Y. Prospective study on late consequences of subclinical non-compliance with immunosuppressive therapy in renal transplant patients. Am J Transplant. 2004 Sep;4(9):1509-13. doi: 10.1111/j.1600-6143.2004.00537.x. PMID 15307839
- [Background] Russell CL, Conn VS, Ashbaugh C, Madsen R, Hayes K, Ross G. Medication adherence patterns in adult renal transplant recipients. Res Nurs Health. 2006 Dec;29(6):521-32. doi: 10.1002/nur.20149. PMID 17131276
- [Background] De Bleser L, Matteson M, Dobbels F, Russell C, De Geest S. Interventions to improve medication-adherence after transplantation: a systematic review. Transpl Int. 2009 Aug;22(8):780-97. doi: 10.1111/j.1432-2277.2009.00881.x. Epub 2009 Apr 6. PMID 19386076
- [Background] Russell C, Conn V, Ashbaugh C, Madsen R, Wakefield M, Webb A, Coffey D, Peace L. Taking immunosuppressive medications effectively (TIMELink): a pilot randomized controlled trial in adult kidney transplant recipients. Clin Transplant. 2011 Nov-Dec;25(6):864-70. doi: 10.1111/j.1399-0012.2010.01358.x. Epub 2010 Nov 16. PMID 21077956
- [Background] Denhaerynck K, Dobbels F, Cleemput I, Desmyttere A, Schafer-Keller P, Schaub S, De Geest S. Prevalence, consequences, and determinants of nonadherence in adult renal transplant patients: a literature review. Transpl Int. 2005 Oct;18(10):1121-33. doi: 10.1111/j.1432-2277.2005.00176.x. PMID 16162098
- [Background] Mange KC, Cizman B, Joffe M, Feldman HI. Arterial hypertension and renal allograft survival. JAMA. 2000 Feb 2;283(5):633-8. doi: 10.1001/jama.283.5.633. PMID 10665703
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] McGillicuddy JW, Gregoski MJ, Weiland AK, Rock RA, Brunner-Jackson BM, Patel SK, Thomas BS, Taber DJ, Chavin KD, Baliga PK, Treiber FA. Mobile Health Medication Adherence and Blood Pressure Control in Renal Transplant Recipients: A Proof-of-Concept Randomized Controlled Trial. JMIR Res Protoc. 2013 Sep 4;2(2):e32. doi: 10.2196/resprot.2633. PMID 24004517